CLINICAL TRIAL: NCT00223938
Title: A Multi-center, Open-label, Randomized, Parallel Group Study of the Efficacy and Safety of Ferrlecit in the Maintenance of Iron Stores and Serum Hemoglobin Concentration in Hemodialysis Patients Receiving Erythropoietin.
Brief Title: Study of the Efficacy and Safety of Ferrlecit in the Maintenance Dosing in Hemodialysis Patients.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated because of significant enrollment challenges
Sponsor: Sanofi (Industry)
Responsible Party: Gary Hoel PhD Executive Director, Watson
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR02023
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Iron; ferrous sulfate; ferric gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Oral Iron
  Interventions: Drug: Oral Iron
- 2 (Experimental): sodium ferric gluconate
  Interventions: Drug: sodium ferric gluconate
- 3 (Experimental): sodium ferric gluconate
  Interventions: Drug: sodium ferric gluconate

INTERVENTIONS:
Drug: Oral Iron — Oral Iron
  Other Names: Ferrous sulfate
  Arms: 1
Drug: sodium ferric gluconate — weekly intravenous injection Dose 1
  Other Names: Ferrlecit
  Arms: 2
Drug: sodium ferric gluconate — weekly intravenous injection Dose 2
  Other Names: Ferrlecit
  Arms: 3

SUMMARY:
This is a phase 4 clinical investigation of the efficacy and safety of Ferrlecit in the maintenance of iron stores and serum hemoglobin concentration in hemodialysis patients receiving Erythropoietin.

DETAILED DESCRIPTION:
A Multi-Center, Open-Label, Parallel Group Study of the efficacy and safety of Ferrlecit in the Maintenance of Iron Stores and Serum Hemoglobin Concentration in Hemodialysis Patients Receiving Erythropoietin. Patients with normal iron indices receive one of two doses of Ferrlecit administered weekly throughout the treatment period. Efficacy was assesses at designated timepoints throughout the study and after the last Ferrlecit dose.

ELIGIBILITY:
Inclusion Criteria:

* Male of female, 18 years old or older.
* Have been receiving chronic hemodialysis therapy
* On stable EPO dosing regimen.
* Have signed patient informed consent.
* Predetermined serum ferritin and TSAT levels.
* Clinical instability - inability to achieve adequate dialysis, abnormal serum albumin and serum glucose.
* Pregnant or lactating.
* A known sensitivity to Ferrlecit

Exclusion Criteria:

* Scheduled for renal transplant.
* A serious concomitant medical disorders incompatible with participation in the study.
* Unable to cooperate or comply with the protocol.
* Use of any investigation agent within 30 days prior to study or during the course of the study.
* Judged by the investigator as unsuitable for enrollment for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2003-12-30 (Actual); Primary Completion 2007-04-27 (Actual); Study Completion 2007-04-27 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the efficacy of two dose levels of Ferrlecit when compared with oral iron when administered as maintenance therapy in iron-replete hemodialysis patients who are receiving Erythropoietin. | 22 weeks

SECONDARY OUTCOMES:
The secondary objectives of this study include comparisons between Ferrlecit treatments to oral iron regarding changes from baseline in hematological parameters, iron indices, EPO requirements and safety. | 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hoel, RPh, PhD, Study Director — Watson Pharmaceuticals
Locations (8):
- United States (8):
  - Hot Springs, Arkansas
  - Orange County, California
  - Simi Valley, California
  - Pembroke Pines, Florida
  - Winston-Salem, North Carolina
  - Canton, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania